CLINICAL TRIAL: NCT00477399
Title: Effect of Four Years Intensive- Versus Regular Follow up, After a One Year Weight Loss Period, in Patients With Morbid Obesity.
Brief Title: Long Term Follow up After 1 Year Initial Lifestyle Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment of study participants
Sponsor: Tor-Ivar Karlsen (Other)
Collaborators: Sykehuset i Vestfold HF (Other)
Responsible Party: Sponsor-Investigator, Tor-Ivar Karlsen, RN PhD, Evjeklinikken
Organization: Evjeklinikken (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK0701
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Obesity; Weight loss maintenance; QOL; Life Style; Follow Up
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): Receiving active follow up (two yearly 1 week stays, telephone follow up, GP-visits)
  Interventions: Behavioral: Long term follow up after intensive lifestyle intervention
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Long term follow up after intensive lifestyle intervention
  Arms: Intervention

SUMMARY:
The effect of non-surgical methods for obesity treatment are not fully documented. This study focus on the long term effect of an intensiv follow up (the "Evje Model") compared to a regular follow up.

The "Evje Model" is a combined model, consisting of repeated stays at a specialist centre, telephone follow up at home, home groups, self monitoring and close contact with the patients' local physician.

DETAILED DESCRIPTION:
200 patients will undergo a 1 year intensive lifestyle intervention.This group will be randomised into an intervention group (n=100) and a control group (n=100). The intervention group will undergo four years of further follow up in accordance with the intervention model, which means two one weeks stays each year at the Evje Clinic, telephone follow up, self monitoring and collaboration with the patients' local physician.

The control group will be followed up by the patients local physician and a yearly control at the Center for Morbid Obesity at Vestfold Hospital (Sykehuset i Vestfold HF).

The purpose is to measure the effect of these two follow up models in regard to weight loss maintanance, Quality of Life and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients, referred from Public Hospitals, with morbid obesity that have undergone one year intensive life style intervention in accordance with the Evje Model.

Exclusion Criteria:

* Pregnancy, major and active psychiatric disease, active and serious eating disorder

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05 (Estimated); Primary Completion 2015-03 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 03.2015

SECONDARY OUTCOMES:
Health related quality of life | 03.2015
Anthropometrics | 03.2015

CONTACTS AND LOCATIONS:
Overall Officials: Joran Hjelmesath, Dr. Med., Study Chair — Sykehuset i Vestfold HF
Locations (1):
- Evjeklinikken AS, Evje, Evjemoen, Norway

REFERENCES:
- [Derived] Karlsen TI, Sohagen M, Hjelmesaeth J. Predictors of weight loss after an intensive lifestyle intervention program in obese patients: a 1-year prospective cohort study. Health Qual Life Outcomes. 2013 Oct 3;11:165. doi: 10.1186/1477-7525-11-165. PMID 24090083
- See also: Home page of Evjeklinikken — http://www.evjeklinikken.no